CLINICAL TRIAL: NCT06527183
Title: Fibromyalgia and Small Fiber Neuropathy : Which Prevalence and Which Relationship With Pain ?
Brief Title: Fibromyalgia and Small Fiber Neuropathy
Acronym: FIBRO-NEP
Status: Recruiting | Type: Observational
Sponsor: Hospital Ambroise Paré Paris (Other)
Responsible Party: Principal Investigator, Nadine ATTAL, Coordinator, Hospital Ambroise Paré Paris
Other Study IDs: 2020-A03400-39
Record Dates: First submitted 2024-07-24; First posted 2024-07-30 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pain Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patients with fibromyalgia: Patients with fibromyalgia based on ACR criteria
  Interventions: Diagnostic Test: Skin punch biopsy to demonstrate small fiber neuropathy
- Patients with other chronic pain (paired for the other groups): Patients with chronic pain other than fibromyalgia and neuropathic pain, eg nociplastic pains or nociceptive pains
  Interventions: Diagnostic Test: Skin punch biopsy to demonstrate small fiber neuropathy
- Paired healthy subjects: Healthy subjects paired for gender and age
  Interventions: Diagnostic Test: Skin punch biopsy to demonstrate small fiber neuropathy

INTERVENTIONS:
Diagnostic Test: Skin punch biopsy to demonstrate small fiber neuropathy — Skin punch biopsy to assess intrapidermal nerve fiber density
  Other Names: Other diagnostic tests will include laser evoked potentiels, quantitative sensory testing, sudoscan, and confocal corneal microscopu

SUMMARY:
The primary objective of this study will be to assess the proportion of fibromyalgia patients with diffuse small-fiber neuropathy (i.e. in the upper and lower limbs) and compare this proportion to patients with other chronic pains (nociplastic, nociceptive) and with healthy controls. Our analysis will be based on the demonstration of structural abnormalities of small nerve fibers by means of skin biopsy, but also of functional abnormalities using four validated tests commonly used in this field: quantitative sensory testing (QST), laser evoked potential recordings, Sudoscan and confocal corneal microscopy. It will thus be possible to verify whether or not patients with small fiber neuropathy have a particular clinical profile in terms of pain, physical activity, comorbidities or pain impact.

DETAILED DESCRIPTION:
Small fiber neuropathy has been observed in a large proportion of fibromyalgia patients. However, the pathophysiological role of these neurological abnormalities in determining the pain and other symptoms of fibromyalgia, and the specificity of these abnormalities, are not well understood.

The primary objective of this study will be to assess the proportion of fibromyalgia patients with diffuse small-fiber neuropathy (i.e. in the upper and lower limbs) and compare this proportion to patients with other chronic pains (nociplastic, nociceptive) and with healthy controls. Our analysis will be based on the demonstration of structural abnormalities of small nerve fibers by means of skin biopsy, but also of functional abnormalities using four validated tests commonly used in this field: quantitative sensory testing (QST), laser evoked potential recordings, Sudoscan and confocal corneal microscopy. It will thus be possible to verify whether or not patients with small fiber neuropathy have a particular clinical profile in terms of pain, physical activity, comorbidities or pain impact.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age with no age limit -
* having given their signed consent to take part in the study
* affiliated to the French social security system
* able to be followed for the entire duration of the study
* reading and understanding French
* accepting the principle of the study and able to comply with its conditions
* suffering from chronic pain for at least six months of at least moderate intensity (≥ 4/10)
* fibromyalgia detected by the FiRST questionnare and defined by the revised diagnostic criteria of the WHO or chronic nociceptive or nociplastic pain without associated fibromyalgia.
* chronic pain for at least 6 months of at least moderate intensity (≥ 4/10)
* untreated or with stable analgesic treatment for at least 2 weeks prior to inclusion- normal neurological examination at inclusion

Exclusion Criteria:

* litigation or compensation-seeking
* cancer for less than 2 years
* known cause of small-fiber neuropathy such as diabetes, systemic disease, hypothyroidism, alcohol, renal failure, genetic disease
* clinical or EMG neuropathy
* peripheral or central nervous system pathology with or without associated neuropathic pain
* uncontrolled chronic pathology such as : morbid obesity, sleep apnea, uncontrolled hypertension, etc. - psychosis, previous suicide attempt
* drug or psychoactive substance abuse
* cognitive or psychological disorders incompatible with compliance with and/or understanding of the protocol
* participation in another biomedical research protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with fibromyalgia, other chronic pains (nociplastic or nociceptive) and healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Prevalence of small fiber neuropathy or pathology as assessed with skin punch biopsy in patients with fibromyalgia as compared to patients with other chronic pains and healthy subjects | Baseline and at 6 months
  intraepidermal nerve fiber density

SECONDARY OUTCOMES:
Correlation between intraepidermal nerve fiber density and pain or other patient reported outcome measures (quality of life, distress, disability...) | Baseline and at 6 months
  Correlation statistics (Spearman Rho)
Investigate the potential specificity of the results obtained by comparing them with pain patients without fibromyalgia or nerve damage (patients with any nociceptive or nociplastic pain without fibromyalgia) matched for age and gender | Baseline and at 6 months
  Direct group comparisons
Monitor the evolution of abnormalities obtained over time (6 months) and correlate them with the evolution of pain and associated symptoms. | 6 months
  Comparison of intraepidermal nerve fiber density and other diagnostic measures between baseline and 6 months
Determine the sensitivity and diagnostic value of corneal confocal microscopy and laser evoked potentials as compared with skin punch biopsy for exploring nociceptive fibers | Baseline and at 6 months
  Sensitivity and specificy of these tests compared to skin punch biopsy
Determine the diagnostic value of the sudoscan and quantified sensory tests compared with other tests for exploring nociceptive fibers in these patients | Baseline and at 6 months
  Sensitivity and specificy of sudoscan and quantitative sensory testing compared to skin punch biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Nadine ATTAL, MD PhD, Principal Investigator — APHP
Locations (2):
- France (2):
  - Inserm U987, Boulogne-Billancourt
  - Centre d'Evaluation et de Traitement de la douleur, Paris

IPD SHARING:
Plan to Share IPD: Undecided